CLINICAL TRIAL: NCT00980629
Title: A Randomized, Placebo-Controlled, Double-blind, Parallel Group, Multi-centre Phase II Dose-Finding Study of M516102 in the Treatment of Pruritus Associated With Atopic Dermatitis
Brief Title: Dose-Finding Study of M516102 in the Treatment of Pruritus Associated With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Allocation: Randomized | Masking: Double
Other Study IDs: M516102-EU03
Record Dates: First submitted 2009-07-24; First posted 2009-09-21 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

INTERVENTIONS:
Drug: M516102 — Twice a day
Drug: placebo — Twice a day

SUMMARY:
This study is to investigate the efficacy and safety of M516102 and to evaluate the dose response relationship of M516102 and placebo, in the treatment of pruritus associated with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients (aged 18-65 years) with a diagnosis of AD.
2. Female patients of child bearing potential must be using a medically acceptable form of contraception.
3. Patients who are able and willing to give signed informed consent.
4. Patients who have pruritus exceed the reference range.

Exclusion Criteria:

1. Patients who have a history of allergy to hydrocortisone.
2. Patients who have a history of relevant drug hypersensitivity.
3. Patients who have a history of contact dermatitis induced by a topical steroid.
4. Patients who are taking, and who are unwilling not to take, any medications or therapy prohibited by the protocol for the complete duration of the study.
5. Patients who have a history or presence of any cancer.
6. Patients who have any renal or liver insufficiency, or clinically significant cardiac, renal or hepatic disease.
7. Patients who, in the opinion of the investigator, are not deemed eligible as determined by medical history, physical examination or clinical laboratory safety tests.
8. Patients who have pruritus associated with conditions other than AD.
9. Patients who have pruritus only on the face and head.
10. Patients who, in the opinion of the investigator, have clinically relevant history or presence of any disease, or surgical history other than AD which is likely to affect the conduct of the study.
11. Patients who have used M5161(active ingredient of M516102).
12. Patients who cannot communicate reliably with the investigator.
13. Patients who are pregnant or lactating.
14. Patients who have used any IMP and/or participated in any clinical trial within 3 months.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2008-08; Study Completion 2010-09

PRIMARY OUTCOMES:
Pruritus score

CONTACTS AND LOCATIONS:
Locations (4):
- Hôpital Morvan, Brest, France
- Universitätsklinikum Münster, Münster, Germany
- Samodzielny Publiczny Szpital Kliniczny Nr 1, Warsaw, Poland
- The Royal Infirmary of Edinburgh, Edinburgh, United Kingdom